CLINICAL TRIAL: NCT02943564
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study of Rapastinel as Adjunctive Therapy in Major Depressive Disorder
Brief Title: A Study of Rapastinel as Adjunctive Therapy in Major Depressive Disorder (RAP-MD-02)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Naurex, Inc, an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAP-MD-02
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Results first posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — GLYX-13 peptide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rapastinel 225 mg (Experimental): Rapastinel 225 milligram (mg) weekly intravenous (IV) injections. Each participant will continue to take the same dose of antidepressant therapy the participant was receiving prior to entering this study throughout treatment.
  Interventions: Drug: Rapastinel
- Rapastinel 450 mg (Experimental): Rapastinel 450 mg weekly IV injections. Each participant will continue to take the same dose of antidepressant therapy the participant was receiving prior to entering this study throughout treatment.
  Interventions: Drug: Rapastinel
- Placebo (Placebo Comparator): Placebo-matching rapastinel weekly IV injections. Each participant will continue to take the same dose of antidepressant therapy the participant was receiving prior to entering this study throughout treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapastinel — Rapastinel pre-filled syringes for weekly IV injections.
  Arms: Rapastinel 225 mg; Rapastinel 450 mg
Drug: Placebo — Placebo-matching rapastinel pre-filled syringes for weekly IV injections.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety, and tolerability of two doses of rapastinel, 225 milligrams (mg) and 450 mg, compared to placebo adjunctive to antidepressant therapy (ADT) in patients with major depressive disorder (MDD) who have a partial response to ADT.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for MDD
* Current major depressive episode of at least 8 weeks and not exceeding 18 months in duration at Visit 1
* Have no more than partial response (< 50% improvement) to ongoing treatment with a protocol-allowed antidepressant
* If female of childbearing potential, have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test.

Exclusion Criteria:

* DSM-5-based diagnosis of any disorder other than MDD that was the primary focus of treatment within 6 months before Visit 1
* Lifetime history of meeting DSM-5 criteria for:

  1. Schizophrenia spectrum or other psychotic disorder
  2. Bipolar or related disorder
  3. Major neurocognitive disorder
  4. Neurodevelopmental disorder of greater than mild severity or of a severity that impacts the participant's ability to consent, follow study directions, or otherwise safely participate in the study
  5. Dissociative disorder
  6. Posttraumatic stress disorder
  7. MDD with psychotic features
* Significant suicide risk, as judged by the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Hoogerheyde, Study Director — Allergan
Locations (66):
- United States (66):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona Department of Psychiatry, Tucson, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - California Pharmaceutical Research Institute, Inc, Anaheim, California
  - ProScience Research Group, Culver City, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Synergy Clinical Research Center of Escondido, Lemon Grove, California
  - Pacific Research Partners; LLC., Oakland, California
  - CITrials, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - PCSD Feighner Research, San Diego, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Reliable Clinical Research, Hialeah, Florida
  - Advanced Research Institute of Miami, Homestead, Florida
  - Innovative Clinical Research, Inc, Lauderhill, Florida
  - International Research Associates, LLC, Miami, Florida
  - Sarkis Clinical Trials, Ocala, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Millenia Psychiatry & Research, Inc, Orlando, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - IRIS Research, Smyrna, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - Phoenix Medical Research, Prairie Village, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - J Gary Booker, MD APMC, Shreveport, Louisiana
  - Pharmasite Research, Inc, Baltimore, Maryland
  - CBH Health, Rockville, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices & Research, Inc., Methuen, Massachusetts
  - BTC of New Bedford, New Bedford, Massachusetts
  - Coastal Research Associates, Weymouth, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - Millennium Psychiatric Associates, Olivette, Missouri
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Pharmaceutical Research Associates Inc, Marlton, New Jersey
  - The Medical Research Network, LLC, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Richard H. Weisler, MD, PA, Raleigh, North Carolina
  - Patient Priority Clinical Site, LLC, Cincinnati, Ohio
  - The Ohio State University Department of Psychiatry, Columbus, Ohio
  - Charak Clinical Research Center, Garfield Heights, Ohio
  - Lindner Center of Hope, Mason, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - Red River Medical Research Center, LLC, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Inc, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - Community Clinical Research, Inc., Austin, Texas
  - BioBehavioral Research of Austin, Austin, Texas
  - Relaro Medical Trials, Dallas, Texas
  - El Campo Clinical Trials, El Campo, Texas
  - Earle Research, Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Family Psychiatry of The Wood, The Woodlands, Texas
  - PRA Health Sciences, Salt Lake City, Utah
  - Pacific Institute of Medical Sciences, Bothell, Washington
  - Eastside Therapeutic Resource, Everett, Washington

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://www.AllerganClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 658 total enrolled. 20 discontinued prior to randomization.
Pre-assignment Details: Prior to randomization, patients entered a 1-wk, double-blind, placebo lead-in period to identify placebo responders. Upon completion of the placebo lead-in period, patients were randomized in 1:1 ratio to receive either rapastinel or placebo. Randomization was stratified by patient's responder status (placebo non-responder vs. placebo responder).
Period: Overall Study
Arm/Group | Placebo | Rapastinel 225 mg | Rapastinel 450 mg
Started | 217 | 211 | 210
Responder | 83 | 77 | 77
Non-Responder | 134 | 134 | 133
Completed | 207 | 198 | 201
Not Completed | 10 | 13 | 9
Not completed — Miscellaneous Reasons | 0 | 0 | 3
Not completed — Site terminated by sponsor | 0 | 1 | 0
Not completed — Non-compliance with study drug | 0 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Protocol Violation | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 5 | 2
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The modified Intent-to-Treat (mITT) Population will consist of all patients who were randomized, received at least 1 dose of IP during the randomized treatment period, and had at least 1 post-randomization assessment of the MADRS total score.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rapastinel 225 mg | Rapastinel 450 mg | Total
Number analyzed (Participants) | 217 | 211 | 210 | 638
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (11.75) | 44.3 (13.16) | 44.7 (12.27) | 44.3 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 147 | 153 | 441
  Male | 76 | 64 | 57 | 197
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 22 | 26 | 73
  Not Hispanic or Latino | 192 | 189 | 184 | 565
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 170 | 162 | 159 | 491
  Black or African American | 41 | 46 | 42 | 129
  Asian | 3 | 1 | 5 | 9
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Multiple | 1 | 1 | 1 | 3
MADRS total score at baseline [Mean (Standard Deviation); unit: Scores on a Scale] — The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement.
  Scores on a Scale | 33.6 (4.47) | 33.5 (4.67) | 33.5 (4.85) | 33.6 (4.70)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at the End of Study
Description: The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement.
Time Frame: Baseline and 3 Weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Rapastinel 225 mg | Rapastinel 450 mg
Number analyzed (Participants) | 217 | 211 | 210
Score on a Scale | -4.9 (0.59) | -4.8 (0.60) | -5.4 (0.60)
Statistical Analysis 1: Comparison: Placebo vs Rapastinel 225 mg; Test type: Superiority; p = 0.8862, Mixed Model Repeated Measures (MMRM); Least Squares Mean Difference = 0.1, 95% CI 2-sided [-1.50 to 1.73]
Statistical Analysis 2: Comparison: Rapastinel 225 mg vs Rapastinel 450 mg; Test type: Superiority; p = 0.5772, Mixed Model Repeated Measures (MMRM); Least Squares Mean Difference = -0.5, 95% CI 2-sided [-2.07 to 1.16]

2. Secondary Outcome: Change From Baseline in MADRS Total Score
Description: as for outcome 1
Time Frame: Baseline and Day 8
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Placebo | Rapastinel 225 mg | Rapastinel 450 mg
Number analyzed (Participants) | 217 | 211 | 210
Score on a Scale | -4.5 (0.51) | -4.6 (0.52) | -4.5 (0.52)
Statistical Analysis 1: Comparison: Placebo vs Rapastinel 225 mg; Test type: Superiority; p = 0.8967, Mixed Model Repeated Measures (MMRM); Least Squares Mean Difference = -0.1, 95% CI 2-sided [-1.48 to 1.29]
Statistical Analysis 2: Comparison: Rapastinel 225 mg vs Rapastinel 450 mg; Test type: Superiority; p = 0.9963, Mixed Model Repeated Measures (MMRM); Least Squares Mean Difference = 0.0, 95% CI 2-sided [-1.38 to 1.39]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for up to 28 days.
Description: The Safety Population will consist of all patients who were randomized and received at least 1 dose of IP during the randomized treatment period.
Arm/Group | Placebo | Rapastinel 225 mg | Rapastinel 450 mg
All-Cause Mortality (participants affected / at risk) | 0/217 | 0/211 | 0/210
Serious Adverse Events (participants affected / at risk) | 1/217 | 1/211 | 1/210
Other Adverse Events (participants affected / at risk) | 14/217 | 11/211 | 14/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=217) | Rapastinel 225 mg (N=211) | Rapastinel 450 mg (N=210)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=217) | Rapastinel 225 mg (N=211) | Rapastinel 450 mg (N=210)
Headache (Nervous system disorders) | 14 | 11 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT02943564/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT02943564/SAP_001.pdf